CLINICAL TRIAL: NCT01215149
Title: A Phase 1 Placebo-controlled, Double-blind, Randomized Trial to Evaluate the Safety and Immunogenicity of Ad26-ENVA and Ad35-ENV HIV Vaccines in Healthy HIV-uninfected Adult Volunteers
Brief Title: Safety and Immunogenicity Study of Ad26-ENVA and Ad35-ENV HIV Vaccines in Healthy HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: HIV Vaccine Trials Network (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Beth Israel Deaconess Medical Center (Other); Ragon Institute of MGH, MIT and Harvard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI B003/ IPCAVD-004
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Group A (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad35-ENV at Month 6. Vaccine:Placebo=10:3
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group B (Experimental): Ad35-ENVA at Month 0 followed by Ad26.ENVA.01 at Month 6. Vaccine:Placebo=10:3
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group C (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad35-ENV at Month 3. Vaccine:Placebo=10:3
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group D (Experimental): Ad35-ENV at Month 0 followed by Ad26.ENVA.01 at Month 3. Vaccine:Placebo=10:3
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group E (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad35-ENV at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group F (Experimental): Ad35-ENV at Month 0 followed by Ad26.ENVA.01 at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group G (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad26.ENVA.01 at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group H (Experimental): Ad35-ENV at Month 0 followed by Ad35-ENV at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Placebo Control
- Group I (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad35-ENV at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group J (Experimental): Ad35-ENV at Month 0 followed by Ad26.ENVA.01 at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group K (Experimental): Ad26.ENVA.01 at Month 0 followed by Ad26.ENVA.01 at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad26.ENVA.01 vaccine; Biological: Placebo Control
- Group L (Experimental): Ad35-ENV at Month 0 followed by Ad35-ENV at Month 3. Vaccine:Placebo=16:4
  Interventions: Biological: Ad35-ENV vaccine; Biological: Placebo Control

INTERVENTIONS:
Biological: Ad35-ENV vaccine — Recombinant adenovirus serotype 35 vector vaccine 5x10^10 vp, delivered IM
  Arms: Group A; Group B; Group C; Group D; Group E; Group F; Group H; Group I; Group J; Group L
Biological: Ad26.ENVA.01 vaccine — Recombinant adenovirus serotype 26 vector vaccine, 5x10^10 vp delivered IM
  Arms: Group A; Group B; Group C; Group D; Group E; Group F; Group G; Group I; Group J; Group K
Biological: Placebo Control — Colorless 10mm Tris/HCl buffer

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Ad26.ENVA.01 and Ad35-ENV in low-risk for HIV-uninfected healthy adults administered in heterologous and homologous prime-boost regimens at different time intervals.

DETAILED DESCRIPTION:
The study is a randomized, double-blind placebo-controlled trial assessing the order of vector priming and boosting (Ad26 versus Ad35), the timing of boost (3 versus 6 months) and the homologous versus heterologous regimen at the 3-month time interval. Groups A-D will be enrolled in Boston, MA, USA, Groups E-H will be enrolled at the East African Clinical Research Centres and Groups I-L will be enrolled at the South African Clinical Research Centres.

Volunteers will be screened up to 56 days before vaccination and will be followed for 12 months after the second vaccination.

Approximately 212 volunteers will be randomized to receive either vaccine or placebo within a group (A-L); Groups A-D, Groups E-H and Groups I-L will be randomized separately. Up to 7% over-enrolment (approximately 15 volunteers) will be allowed to facilitate enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, as assessed by a medical history, physical exam, and laboratory tests;
* At least 18 years of age on the day of screening and has not reached his/her 51st birthday on the day of first vaccination;
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study;
* In the opinion of the Principal Investigator or designee, and based on Assessment of Informed Consent Understanding (AOU) results, has understood the information provided and potential risks linked to vaccination and participation in the trial; written informed consent will be provided by the volunteer before any study-related procedures are performed;
* Willing to undergo HIV testing, risk reduction counselling, receive HIV test results and committed to maintaining low risk behaviour for the trial duration as defined by the protocol;
* If a female of childbearing potential, willing to use an effective non-barrier method of contraception (oral or injectable hormonal contraceptive; intrauterine device [IUD]) from screening until at least 4 months after the last study vaccination;
* Assessed by the clinic staff as being at "low risk" for HIV infection on the basis of sexual behaviours within the 12 months prior to enrolment;
* All female volunteers must be willing to undergo pregnancy tests at time points indicated in the protocol and must test negative prior to each study vaccination;
* All sexually active males (unless anatomically sterile) must be willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until at least 4 months after the last vaccination;
* Willing to forgo donations of blood or any other tissues during the study and, for those who test HIV positive due to trial vaccination (vaccine-induced HIV seropositivity), until the anti-HIV antibody titers become undetectable.

Exclusion Criteria

* Confirmed HIV-1 or HIV-2 infection;
* Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted); immunosuppressive, anticancer, antituberculosis or other medications considered significant by the investigator within the previous 6 months;
* Any clinically significant acute or chronic medical condition that is considered progressive, or in the opinion of the investigator, makes the volunteer unsuitable for participation in the study;
* Reported risky behaviour for HIV infection within 12 months prior to vaccination, as defined by the protocol
* If female, pregnant or planning a pregnancy within 4 months after last vaccination; or lactating;
* Asthma requiring high-dose oral or inhaled corticosteroids;
* Fever > 100.4° F/38.0° C within 72 hours prior to vaccine administration;
* Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has IM injections and blood draws without any adverse experience is eligible);
* History of splenectomy;
* Any abnormal laboratory parameters as defined by the protocol;
* Receipt of live-attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with Investigational Product (within 14 days for live attenuated influenza vaccine [LAIV]); or receipt of other vaccine (e.g., influenza, pneumococcal), allergy treatment with antigen injections or tuberculin skin test within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product;
* Receipt of blood transfusion or blood-derived products within the previous 3 months;
* Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study;
* Receipt of another investigational HIV vaccine candidate (Note: receipt of an HIV vaccine control or placebo will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval);
* History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulty, angioedema);
* Confirmed diagnosis of active hepatitis B, hepatitis C or active syphilis;
* Seizure disorder: A participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years.);
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 15-18 months approximately
  To evaluate the safety and tolerability of Ad26.ENVA.01 and Ad35-ENV administered in heterologous and homologous prime-boost regimens.

SECONDARY OUTCOMES:
Immunogenicity | 12 months
  * To evaluate the immunogenicity of Ad26.ENVA.01 and Ad35-ENV administered in heterologous prime-boost regimens at 3 versus 6 month intervals
  * To evaluate the immunogenicity of Ad26.ENVA.01 and Ad35-ENV administered in heterologous and homologous prime-boost regimens at 3 month interval
  * To evaluate anti-vector immunity induced by Ad26.ENVA.01 and Ad35-ENV administered in heterologous and homologous prime-boost regimens

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Principal Investigator — Brigham and Women's Hospital, Boston, MA, USA; Gaudensia Mutua, MB ChB, MPH, Principal Investigator — Kenya AIDS Vaccine Initiative, Kangemi, Kenya; Etienne Karita, MD, M.Sc., MSPH, Principal Investigator — Projet San Francisco; Linda-Gail Bekker, MD, Principal Investigator — Desmond Tutu HIV Foundation-Emavundleni Research Center; Glenda Gray, MBBCH, FCPaeds(SA), Principal Investigator — Perinatal HIV Research Unit; Liesl Page-Shipp, Principal Investigator — Aurum Institute
Locations (6):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- Kenya AIDS Vaccine Initiative, Kangemi, Kenya
- Projet San Francisco, Kigali, Rwanda
- South Africa (3):
  - Desmond Tutu HIV Foundation-Emavundleni Research Centre, Cape Town (Nyanga)
  - Aurum Institute, Klerksdorp
  - Perinatal HIV Research Unit, Soweto

REFERENCES:
- [Derived] Baden LR, Karita E, Mutua G, Bekker LG, Gray G, Page-Shipp L, Walsh SR, Nyombayire J, Anzala O, Roux S, Laher F, Innes C, Seaman MS, Cohen YZ, Peter L, Frahm N, McElrath MJ, Hayes P, Swann E, Grunenberg N, Grazia-Pau M, Weijtens M, Sadoff J, Dally L, Lombardo A, Gilmour J, Cox J, Dolin R, Fast P, Barouch DH, Laufer DS; B003-IPCAVD004-HVTN091 Study Group. Assessment of the Safety and Immunogenicity of 2 Novel Vaccine Platforms for HIV-1 Prevention: A Randomized Trial. Ann Intern Med. 2016 Mar 1;164(5):313-22. doi: 10.7326/M15-0880. Epub 2016 Feb 2. PMID 26833336
- See also: International AIDS Vaccine Initiative — http://www.iavi.org